CLINICAL TRIAL: NCT04960488
Title: Multidisciplinary Collaborative Carotid Endarterectomy and Coronary Artery Bypass Graft Surgery to Optimize the Management of High-risk Patients During the Perioperative Period
Brief Title: Multidisciplinary CAE and CABG Surgery to Optimize the Management of High-risk Patients During the Perioperative Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M2020062
Record Dates: First submitted 2021-07-04; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2019-12

CONDITIONS: Carotid Endarterectomy; Coronary Artery Bypass Grafting
MeSH Terms: interventions — Endarterectomy, Carotid; Coronary Artery Bypass

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- carotid endarterectomy and coronary artery bypass grafting (Experimental): carotid endarterectomy and coronary artery bypass grafting
  Interventions: Procedure: carotid endarterectomy and coronary artery bypass grafting
- carotid endarterectomy (Active Comparator): carotid endarterectomy
  Interventions: Procedure: carotid endarterectomy and coronary artery bypass grafting

INTERVENTIONS:
Procedure: carotid endarterectomy and coronary artery bypass grafting — carotid endarterectomy and coronary artery bypass grafting

SUMMARY:
This project uses concurrent CEA+CABG combined surgery on high-risk patients with severe carotid artery stenosis and severe coronary artery stenosis. After multidisciplinary preoperative evaluation, intraoperative electrophysiological monitoring, and postoperative management standards, compare CEA+CABG combined operations during the same period And the advantages and disadvantages of a single CABG or CEA operation, the purpose is to explore the best surgical treatment plan, establish an interdisciplinary clinical medicine platform centered on patients with heart and cerebrovascular diseases, and develop a standard procedure and The perioperative management is standard, so it is particularly important and naturally has its advanced significance.

DETAILED DESCRIPTION:
This project uses concurrent carotid endarterectomy and coronary artery bypass grafting combined surgery on high-risk patients with severe carotid artery stenosis and severe coronary artery stenosis. After multidisciplinary preoperative evaluation, intraoperative electrophysiological monitoring, and postoperative management standards, compare CEA+CABG combined operations during the same period And the advantages and disadvantages of a single CABG or CEA operation, the purpose is to explore the best surgical treatment plan, establish an interdisciplinary clinical medicine platform centered on patients with heart and cerebrovascular diseases, and develop a standard procedure and The perioperative management is standard, so it is particularly important and naturally has its advanced significance.

ELIGIBILITY:
Inclusion Criteria:

* (1) In patients with symptomatic carotid artery stenosis, the preoperative CTA or DSA, combined with carotid ultrasound and high-resolution magnetic resonance clearly diagnosed the degree of carotid artery stenosis on the responsible side>50%; (2) Patients with asymptomatic carotid artery stenosis before operation CTA or DSA, combined with carotid ultrasound and high-resolution magnetic resonance, clearly diagnosed the carotid artery stenosis rate of the affected side>70%; (3) All patients with carotid artery stenosis were located in the surgically accessible position, without complete carotid artery occlusion or intracranial segment Severe vascular stenosis; (4) The stenosis rate of the left main coronary artery by coronary angiography is more than 70%, or the disease of the three main vessels is more than 50%, and the bridging condition is good.

Exclusion Criteria:(1) The disease is beyond the reach of surgery (such as C2 level or above); (2) The symptoms of hypertension are not effectively controlled before surgery (systolic blood pressure> 180mmHg); (3) Carotid artery stenosis caused by non-atherosclerosis , Such as arteritis, arterial dissection, vascular congenital malformations, etc.; (4) combined with hemorrhagic cerebrovascular diseases such as intracranial aneurysms or vascular malformations; (5) combined with blood system diseases that lead to coagulation dysfunction that cannot be corrected or refused to accept blood and blood Importers of products; (6) Pregnancy or perinatal period.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Cerebral oxygen saturation | Intraoperative
  Cerebral oxygen saturation monitoring

CONTACTS AND LOCATIONS:
Overall Officials: tao wang, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No